CLINICAL TRIAL: NCT00916227
Title: A Study of ARRY-614 in Patients With Low or Intermediate-1 Risk Myelodysplastic Syndrome
Status: Completed | Phase: Phase 1 | Type: Interventional
Sponsor: Array Biopharma, now a wholly owned subsidiary of Pfizer (Industry)
Responsible Party: Sponsor
Organization: Array BioPharma (Industry)
Allocation: Not Applicable | Model: Single Group | Masking: None | Purpose: Treatment
Other Study IDs: ARRAY-614-111
Record Dates: First submitted 2009-06-03; First posted 2009-06-09 (Estimated); Last update posted 2020-09-09 (Actual); Status verified 2020-09

CONDITIONS: Myelodysplastic Syndromes
Keywords: Low or Intermediate-1 Risk Myelodysplastic Syndrome
MeSH Terms: conditions — Myelodysplastic Syndromes | interventions — pexmetinib

ARMS (1):
- ARRY-614 (Experimental)
  Interventions: Drug: ARRY-614, p38/Tie2 inhibitor; oral

INTERVENTIONS:
Drug: ARRY-614, p38/Tie2 inhibitor; oral — Part 1: multiple dose, escalating; Part 2: multiple dose, single schedule.

SUMMARY:
This is a Phase 1 study during which patients with low or intermediate-1 risk myelodysplastic syndrome (MDS) will receive investigational study drug ARRY-614.

This study has 2 parts. In the first part, patients will receive increasing doses of study drug, given either with food or without food, in order to achieve the highest dose of the study drug possible that will not cause unacceptable side effects. Approximately 60 patients from the US will be enrolled in Part 1 (Completed).

In the second part of this study, patients will receive the best dose of study drug, given either with food or without food, determined from the first part of the study and will be followed to see what side effects and effectiveness the study drug has, if any, in treating the cancer. Approximately 40 patients from the US will be enrolled in Part 2 (Completed).

ELIGIBILITY:
Key Inclusion Criteria (Part 1 and Part 2):

* Diagnosis of MDS by bone marrow biopsy.
* International Prognostic Scoring System (IPSS) score of low or intermediate-1 risk MDS.
* May have received prior therapy for MDS.
* Eastern Cooperative Oncology Group (ECOG) performance status (PS) between 0 and 2.
* Adequate liver and renal function.
* Additional criteria exist.

Key Exclusion Criteria (Part 1 and Part 2):

* History of bone marrow transplant.
* Concomitant malignancies or previous malignancies with less than a 2-year disease-free interval at the time of enrollment.
* Treatment with an investigational medicinal product that is not expected to be cleared by the first dose of study drug or that has demonstrated to have late side effects.
* Known positive serology for the human immunodeficiency virus (HIV), hepatitis C and/or active hepatitis B.
* Additional criteria exist.

Min Age: 18 Years | Sex: All | Healthy Volunteers: No
Age Groups: Adult, Older Adult
Enrollment: 45 (Actual)
Dates: Start 2009-06; Primary Completion 2012-01 (Actual)

PRIMARY OUTCOMES:
Characterize the safety profile of the study drug, in either the fasted or fed state, in terms of adverse events, clinical laboratory tests and electrocardiograms. | Part 1, one year; Part 2, one year
Establish the maximum tolerated dose (MTD) of the study drug. | Part 1, one year
Characterize the pharmacokinetics of the study drug and a metabolite under either fasted or fed conditions. | Part 1, one year; Part 2, one year

SECONDARY OUTCOMES:
Assess the efficacy of study drug in terms of response, duration of response and hematologic improvement. | Part 1, one year; Part 2, one year

CONTACTS AND LOCATIONS:
Overall Officials: Pfizer CT.gov Call Center, Study Director — Pfizer
Locations (3):
- United States (3):
  - Moffitt Cancer Center, Tampa, Florida
  - Winship Cancer Institute, Atlanta, Georgia
  - MD Anderson Cancer Center, Houston, Texas